CLINICAL TRIAL: NCT07233395
Title: Comparison of the Effectiveness of Dextrose Prolotherapy and Extracorporeal Shock Wave Therapy (ESWT) in Plantar Fasciitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Zeynep Karakuzu Güngör, Physical Medicine and Rehabilitation, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KanuniSSTRH-PF-2025
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Plantar Fasciitis
Keywords: Dextrose Prolotherapy; Extracorporeal Shock Wave Therapy (ESWT); Physical Medicine and Rehabilitation
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Prolotherapy; Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups. One group will receive dextrose prolotherapy and the other will receive extracorporeal shock wave therapy (ESWT).
  The study aims to compare the effectiveness of these two regenerative treatment methods in patients with plantar fasciitis.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded to treatment allocation. Participants and care providers will be aware of the intervention due to the nature of the treatments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dextrose Prolotherapy (Experimental): Participants in this group will receive dextrose prolotherapy twice, at two-week intervals.
  A 5 mL syringe will be prepared with 2.5 mL of 30% dextrose, 2 mL of isotonic saline, and 0.5 mL of 2% lidocaine (final 15% dextrose solution).
  Injections will be administered into seven points around the plantar fascia origin and insertion under aseptic conditions.
  Interventions: Procedure: Dextrose Prolotherapy
- Extracorporeal Shock Wave Therapy (ESWT) (Active Comparator): Participants in this group will receive extracorporeal shock wave therapy (ESWT) twice per week for a total of four sessions.
  The treatment will be applied to the plantar fascia insertion using a standard clinical ESWT device following manufacturer guidelines.
  Interventions: Device: Extracorporeal Shock Wave Therapy (ESWT)

INTERVENTIONS:
Procedure: Dextrose Prolotherapy — Participants in this group will receive dextrose prolotherapy twice, at two-week intervals.
  A 5 mL syringe containing 2.5 mL of 30% dextrose, 2 mL isotonic saline, and 0.5 mL 2% lidocaine (final 15% dextrose solution) will be injected into seven points around the plantar fascia origin under aseptic conditions.
  Other Names: Prolotherapy Injection
  Arms: Dextrose Prolotherapy
Device: Extracorporeal Shock Wave Therapy (ESWT) — Participants in this group will receive extracorporeal shock wave therapy (ESWT) twice per week for a total of four sessions.
  The treatment will be applied to the plantar fascia insertion area using a standard clinical shock wave therapy device.
  Energy level, frequency, and pulse count will be set according to manufacturer recommendations and standard clinical protocols.
  Other Names: Shock Wave Therapy
  Arms: Extracorporeal Shock Wave Therapy (ESWT)

SUMMARY:
Plantar fasciitis is a degeneration of the plantar aponeurosis and is the most common cause of heel pain (11-15%). Although seen in both sexes, plantar fasciitis is more common in women, usually unilateral and bilateral in 30% of cases . The most widely accepted view regarding the formation of plantar fasciitis is that it is a degenerative process caused by myxoid degeneration, microtears, collagen necrosis, and angiofibroblastic hyperplasia, resulting from repetitive microtrauma to the plantar fascia, particularly at the calcaneal insertion site. It is not inflammatory . The purpose of this study was to compare the effectiveness of prolotherapy, a regenerative treatment, and ESWT in the treatment of plantar fasciitis.

DETAILED DESCRIPTION:
Plantar fasciitis is known as the most common cause of heel pain in adults. While its incidence increases between the ages of 40 and 60, it is more common in runners, those who work in positions requiring prolonged standing, overweight individuals, and those with certain biomechanical foot problems. Diagnosis of plantar fasciitis can be easily made through history and physical examination. Conservative methods are the first line of treatment. Local injections and ESWT are used in patients who fail to improve despite conservative treatment. ESWT and Prolotherapy are treatment methods that induce regeneration by creating a controlled inflammation. This prospective study aims to compare the effectiveness of ESWT and Prolotherapy, which have similar mechanisms of action, in the treatment of plantar fasciitis and to identify the more effective method.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of plantar fasciitis

Ages 18 to 75 years

Both male and female participants

Heel pain localized to the medial calcaneal tubercle for more than 3 months

Morning first-step pain and pain increasing with daily loading

Willingness to participate and provide written informed consent

Patients presenting to Kanuni Sultan Süleyman Training and Research Hospital

Exclusion Criteria:

Cardiac pacemaker

Type 1 or Type 2 diabetes mellitus

History of inflammatory rheumatic disease

Bleeding disorders

Use of anticoagulant medications other than aspirin

Allergy to dextrose

Previous foot or ankle surgery

Peripheral neuropathy

S1 radiculopathy in the same extremity

Local corticosteroid injection to the plantar fascia within the last 3 months

ESWT applied to the plantar fascia within the last 3 months

Physical therapy applied to the foot/ankle in the last 3 months

Cognitive dysfunction

Active infection at the planned injection site

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Change in Heel Pain Intensity (VAS Score) | Baseline, 6 weeks, 12 weeks
  Heel pain intensity will be assessed using a 10-cm Visual Analog Scale (VAS) at baseline, 6 weeks, and 12 weeks. The primary outcome is the change in VAS score from baseline to week 12 in each treatment group.

SECONDARY OUTCOMES:
Change in Foot Function Index (FFI) Total Score | Baseline, 6 weeks, 12 weeks
  Functional status will be assessed using the Foot Function Index (FFI), which evaluates pain, disability, and activity limitation related to foot function. The total FFI score will be recorded at baseline, 6 weeks, and 12 weeks. The secondary outcome is the change in FFI total score over time.
Change in Roles and Maudsley Score | Baseline, 6 weeks, 12 weeks
  The Roles and Maudsley functional pain score will be used to evaluate treatment response. Patients grade their condition on a 4-point scale from "excellent" to "poor." Scores will be obtained at baseline, 6 weeks, and 12 weeks. Improvement in score indicates better clinical outcome.

CONTACTS AND LOCATIONS:
Overall Officials: ZEYNEP KARAKUZU GÜNGÖR, MD, Principal Investigator — Kanuni Sultan Süleyman Training and Research Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. Data will only be accessible to the research team in accordance with institutional ethical guidelines and patient confidentiality regulations.